CLINICAL TRIAL: NCT02631161
Title: Randomized Controlled Trial on Glass Hybrid Versus Composite Restorations of Non-carious Cervical Lesions
Brief Title: Glass Hybrid Versus Composite Restorations of Non-carious Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: GC Europe (Industry)
Responsible Party: Principal Investigator, Falk Schwendicke, PD Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHyComp
Record Dates: First submitted 2015-12-07; First posted 2015-12-16 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Dental Cervical Non-carious Lesion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EQUIA forte (Experimental): Dental non-carious cervical restorations are being restored with a glass hybrid restorative system (Medical product: EQUIA forte).
  Interventions: Other: Equia Forte
- Filtek Supreme XT/Clearfil SE Bond (Active Comparator): Dental non-carious cervical restorations are being restored with a composite resin based material/Adhesive combination (Medical product: Filtek Supreme XT/Clearfil SE Bond).
  Interventions: Other: Filtek Supreme XT/Clearfil SE Bond

INTERVENTIONS:
Other: Equia Forte — Restoration of cavities with a Glasshybrid material (Equia Forte)
  Arms: EQUIA forte
Other: Filtek Supreme XT/Clearfil SE Bond — Restoration of cavities with a composite resin based material after placing an adhesive
  Arms: Filtek Supreme XT/Clearfil SE Bond

SUMMARY:
A glass hybrid restorative system (EQUIA forte) clinically compared to a composite resin based material (Clearfil SE Bond, Filtek Supreme XT) for the treatment of dental non-carious cervical lesions.

DETAILED DESCRIPTION:
This is a prospective, randomized, monocenter parallel group study on restoration of tooth with non-carious cervical restorations. Each patient receives cervical restoration(s) either with glass hybrid EQUIA forte or with composite resin/adhesive combination Filtek Supreme XT/Clearfil SE Bond in anterior/posterior tooth region. Restorations will be provided by one experienced operator. One of two independent examiners will evaluate the restorations at baseline (1 week after placement), and after 18, and 36 months according to the FDI criteria. Reliability of examination will be assessed on a random sample of 30 restorations.

ELIGIBILITY:
Inclusion Criteria:

* indication of a restorative treatment for a sclerotic non-carious cervical lesion
* lesions should be accessible for treatment and visual-tactile re-evaluation
* sufficient moisture control should be possible
* cervical margins should be located in dentin whereas the coronal margin should be located in enamel

Exclusion Criteria:

* allergy/hypersensitivity against any of the used materials
* participants should not be systematically ill, disabled, pregnant or participating in another study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Number of restorations with a re-intervention per all restorations | 36 months
  Number of all restorations with a re-intervention being required per all placed restorations (events/sample)

SECONDARY OUTCOMES:
Restoration score | 36 months
  score according to FDI criteria
Costs for initial and retreatment | recorded initially and, if required, each re-treatment appointment, over the total trial period (i.e. expected 36 months)
  Costs incurred for staff and material for initial and re-treatments

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Paris, Prof. Dr., Study Director — Abteilung für Zahnerhaltung und Präventivzahnmedizin, Charité Berlin
Locations (1):
- Charité Centrum für Zahn-, Mund- und Kieferheilkunde, Abteilung für Zahnerhaltungskunde und Präventivzahnmedizin, Berlin, Germany

REFERENCES:
- [Derived] Gostemeyer G, Seifert T, Jeggle-Engbert LM, Paris S, Schwendicke F. Glass Hybrid Versus Nanocomposite for Restoration of Sclerotic Non-carious Cervical Lesions: 18-Month Results of a Randomized Controlled Trial. J Adhes Dent. 2021 Dec 3;23(6):487-496. doi: 10.3290/j.jad.b2287831. PMID 34817964
- [Derived] Schwendicke F, Muller A, Seifert T, Jeggle-Engbert LM, Paris S, Gostemeyer G. Glass hybrid versus composite for non-carious cervical lesions: Survival, restoration quality and costs in randomized controlled trial after 3 years. J Dent. 2021 Jul;110:103689. doi: 10.1016/j.jdent.2021.103689. Epub 2021 May 9. PMID 33979577